CLINICAL TRIAL: NCT00004786
Title: Phase III Randomized, Double-Blind, Placebo-Controlled Study of Oral Iloprost for Raynaud's Phenomenon Secondary to Systemic Sclerosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: University of Pittsburgh (Other)
Organization: Office of Rare Diseases (ORD) (NIH)
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: 199/11876; UPITTS-951019
Record Dates: First submitted 2000-02-24; First posted 2000-02-25 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2001-12

CONDITIONS: Systemic Sclerosis; Raynaud Disease
Keywords: Raynaud's syndrome; arthritis & connective tissue diseases; cardiovascular and respiratory diseases; rare disease; systemic sclerosis
MeSH Terms: conditions — Scleroderma, Systemic; Raynaud Disease; Arthritis; Connective Tissue Diseases; Respiratory Tract Diseases; Rare Diseases | interventions — Iloprost

INTERVENTIONS:
Drug: iloprost

SUMMARY:
OBJECTIVES:

I. Evaluate the safety and efficacy of oral iloprost, a prostacyclin analog, in patients with Raynaud's phenomenon secondary to systemic sclerosis.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: This is a randomized, double-blind study. Patients are stratified by participating institution and digital cutaneous ulcers.

Patients receive oral iloprost or placebo twice daily for 6 weeks. Thrombolytic drugs, oral anticoagulants, and heparin are prohibited on study. Concurrent therapy with angiotensin-converting enzyme inhibitors for Raynaud's is prohibited; calcium channel blockers for severe digital ischemia are allowed as needed.

Patients are followed at 2 and 6 weeks.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics--

* Raynaud's phenomenon secondary to systemic sclerosis (SS) SS meets American College of Rheumatology diagnostic criteria
* At least 6 Raynaud's attacks per week

--Prior/Concurrent Therapy--

* No prior participation in oral iloprost study
* At least 4 weeks since participation in other investigational drug studies
* At least 2 months since prostanoid therapy
* At least 12 months since sympathectomy of upper limb
* Ongoing therapy for systemic sclerosis may continue on study Raynaud's therapy discontinued at entry

--Patient Characteristics--

Hematopoietic: No platelet disorder

Hepatic: No bleeding diathesis

Renal: Creatinine clearance (estimated) at least 30 mL/min

Cardiovascular:

No unstable angina pectoris

None of the following within 3 months:

* Stroke
* Transient ischemic attack
* Myocardial infarction

Other:

* No active cancer or other uncontrolled disease
* No current history of alcohol or drug abuse
* No mental disorder precluding compliance
* No pregnant or nursing women
* Negative pregnancy test required of fertile women
* Adequate contraception required of fertile women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200
Dates: Start 1995-12

CONTACTS AND LOCATIONS:
Overall Officials: Thomas A. Medsger, Jr., Study Chair — University of Pittsburgh